CLINICAL TRIAL: NCT01474369
Title: A Phase 3, Randomized, Double Blind, Placebo Control, Multicenter Study to Evaluate the Efficacy and Safety of TAK- 438 (10 and 20 mg Once-Daily) in Patients With Non-Erosive Gastroesophageal Reflux Disease.
Brief Title: Efficacy of TAK-438 Compared to Placebo in the Treatment of Non-Erosive Gastroesophageal Reflux Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-438/CCT-201; U1111-1125-1115 (Registry Identifier: WHO); JapicCTI-111663 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2011-10-24; First posted 2011-11-18 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-07

CONDITIONS: Non-erosive Gastroesophageal Reflux Disease
Keywords: Drug Therapy
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- TAK-438 10 mg QD (Experimental)
  Interventions: Drug: TAK-438
- TAK-438 20 mg QD (Experimental)
  Interventions: Drug: TAK-438
- Placebo QD (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TAK-438 — TAK-438 10 mg, tablets, orally, once daily for 4 weeks. Thereafter, TAK-438 placebo tablets, orally, once daily for 1 week.
  Arms: TAK-438 10 mg QD
Drug: TAK-438 — TAK-438 20 mg, tablets, orally, once daily for 4 weeks. Thereafter, TAK-438 placebo tablets, orally, once daily for 1 week.
  Arms: TAK-438 20 mg QD
Drug: Placebo — TAK-438 placebo-matching tablets, orally, once daily for 5 weeks.
  Arms: Placebo QD

SUMMARY:
The purpose of this study is to investigate the superiority of efficacy of TAK-438, once daily (QD), to placebo in patients with non-erosive gastroesophageal reflux disease.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with grade N or M in the modified LA classification system confirmed by endoscopy at initiation of the pre-observation period (VISIT 1).
2. Participants with repeated acid reflux symptoms (heartburn or regurgitation) for 2 days or more in one week in the 3 weeks before initiation of initiation of the pre-observation period (VISIT 1).
3. Participants with severity* of moderate or higher for acid reflux symptoms (heartburn or regurgitation) in the 3 weeks before initiation of the pre-observation period (VISIT 1)

   * Severity: No symptoms, very mild (symptoms present but often forgotten), mild (not so painful), moderate (rather painful), severe (painful) and very severe (painful enough to affect night time sleep or daily activities)
4. Outpatients (hospitalization for testing possible)

Exclusion Criteria:

1. Participants with an esophagus-related complication [Barrett's esophagus (3 cm or more, LSBE), eosinophilic esophagitis, esophageal varices, scleroderma, viral or fungal infections, esophageal stenosis, etc.], or a history of radiotherapy or cryotherapy of the esophagus, a caustic or physiochemical trauma (esophageal sclerotherapy, etc.). However, participants with Barrett's esophagus (less than 3 cm, SSBE) or Schatzki's ring (mucosal tissue ring around inferior esophageal sphincter) are allowed to be included.
2. Participants who have received surgery or treatment affecting gastroesophageal reflux (cardioplasty, dilation of esophageal stenosis [excluding Schatzki's ring], etc.), or who have a history of surgery of stomach or duodenum (excluding removal of benign polyp under endoscopy)
3. Participants who have acute upper gastrointestinal bleeding, gastric ulcers (mucosal defects associated with white coating) or duodenal ulcers (mucosal defect with white coating) within 30 days before initiation of the pre-observation period (VISIT 1) However, participants with gastric or duodenal erosions are allowed to be included.
4. Participants with acute gastritis or acute exacerbation of chronic gastritis as a complication
5. Participants with a previous or current history of the Zollinger-Ellison syndrome or other gastric acid hypersecretion disorders
6. Participants with a history of chest pain due to heart disease or with chest pains suspected of being caused by heart disease within one year before initiation of the pre-observation period (VISIT 1)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 827 (Actual)
Dates: Start 2011-12; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Percentage of symptom-free days of heartburn symptoms | Week 4
  Heartburn symptoms will be collected by participant diaries.
Cumulative symptom improvement rate of heartburn symptoms | Week 4
  Heartburn symptoms will be collected by participant diaries.
Severity of heartburn symptoms | Week 4
  Heartburn symptoms will be collected by participant diaries.

SECONDARY OUTCOMES:
Heartburn symptoms stratified by response (improvement or non-improvement) at Week 2 | Week 4
  Heartburn symptoms will be collected by participant diaries. Percentage of symptom-free days, cumulative symptom improvement rate, and severity of heartburn symptoms are evaluation parameters.
Heartburn Symptoms Stratified by Baseline Endoscopic Findings (Grade N or M) | Week 4
  Heartburn symptoms collected by participant diaries. Percentage of symptom-free days, cumulative symptom improvement rate and severity of heartburn symptoms=evaluation parameters. Participants with Non-Erosive Gastroesophageal Reflux Disease divided into Grade N (endoscopically normal) and M (minimal change) by modified Los Angeles Classification System. Grade definitions: Grade N (endoscopically normal), M (minimal change), A (Mucosal break <5 mm) B (Mucosal break ≥5 mm) C (Mucosal break continuous between 2 or more folds and <75% of circumference) and D (Mucosal break ≥75% of circumference).
Heartburn symptoms stratified by combination of response at Week 2 and baseline endoscopic findings (improvement and grade N, improvement and grade M, non-improvement and grade N, non-improvement and grade M.) | Week 4
  Heartburn symptoms will be collected by participant diaries. Percentage of symptom-free days, cumulative symptom improvement rate, and severity of heartburn symptoms are evaluation parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Senior Manager, Study Director — Takeda
Locations (52):
- Japan (52):
  - Nagoya, Aichi-ken
  - Abiko-shi, Chiba
  - Kashiwa-shi, Chiba
  - Noda, Chiba
  - Yachiyo-shi, Chiba
  - Saijo-shi, Ehime
  - Fukuoka, Fukuoka
  - Itoshima-shi, Fukuoka
  - Kasuya-gun, Fukuoka
  - Onga-gun, Fukuoka
  - Kouriyama-shi, Fukushima
  - Gifu, Gifu
  - Takayama-shi, Gifu
  - Annaka-shi, Gunma
  - Hiroshima, Hiroshima
  - Asahikawa-shi, Hokkaido
  - Sapporo, Hokkaido
  - Amagasaki-shi, Hyōgo
  - Kobe, Hyōgo
  - Nishinomiya-shi, Hyōgo
  - Takarazuka-shi, Hyōgo
  - Sagamihara-shi, Kanagawa
  - Yokohama, Kanagawa
  - Kochi, Kochi
  - Suzaki-shi, Kochi
  - Kumamoto, Kumamoto
  - Kyoto, Kyoto
  - Sendai, Miyagi
  - Nagasaki, Nagasaki
  - Ōita, Oita Prefecture
  - Okayama, Okayama-ken
  - Osaka, Osaka
  - Takatsuki-shi, Osaka
  - Saga, Saga-ken
  - Kumagaya-shi, Saitama
  - Saitama-shi, Saitama
  - Tokorozawa-shi, Saitama
  - Otawara-shi, Tochigi
  - Bunkyo-ku, Tokyo
  - Chiyoda-ku, Tokyo
  - Chuo-ku, Tokyo
  - Hachioji-shi, Tokyo
  - Kokubunji-shi, Tokyo
  - Nakano-ku, Tokyo
  - Oota-ku, Tokyo
  - Setagaya-ku, Tokyo
  - Shibuya-ku, Tokyo
  - Shinjuku-ku, Tokyo
  - Shimonoseki-shi, Yamaguchi
  - Kofu, Yamanashi
  - Turu-shi, Yamanashi
  - Yamagata, Ymagata

REFERENCES:
- [Derived] Kinoshita Y, Sakurai Y, Shiino M, Kudou K, Nishimura A, Miyagi T, Iwakiri K, Umegaki E, Ashida K. Evaluation of the Efficacy and Safety of Vonoprazan in Patients with Nonerosive Gastroesophageal Reflux Disease: A Phase III, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study. Curr Ther Res Clin Exp. 2016 Dec 21;81-82:1-7. doi: 10.1016/j.curtheres.2016.12.001. eCollection 2016. PMID 28119763